CLINICAL TRIAL: NCT06603948
Title: Colorectal Adenoma Detection Using Spectral Focused Imaging Versus White Light Imaging: a Parallel Randomized Controlled Trial
Brief Title: Spectral Focused Imaging Versus White Light Imaging in Colorectal Adenoma Detection
Acronym: SFI verus WLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: First Affiliated Hospital of Ningbo University (Network); Nanchong Central Hospital (Other Government); First Affiliated Hospital of Xinjiang Medical University (Other); West China Forth Hospital (Unknown); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Seventh Medical Center of PLA Army General Hospital (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: LY2024-136-C
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Adenoma
Keywords: Spectral Focused Imaging; Colorectal adenoma; ADR

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SFI (Experimental): Spectral Focused Imaging
  Interventions: Device: Spectral Focused Imaging
- WLI (Placebo Comparator): White Light Imaging
  Interventions: Device: White Light Imaging

INTERVENTIONS:
Device: Spectral Focused Imaging — Use of SFI for colon inspection during both insertion and withdrawal phase of colonoscopy
  Arms: SFI
Device: White Light Imaging — Use of WLI for colon inspection during both insertion and withdrawal phase of colonoscopy
  Arms: WLI

SUMMARY:
Spectral Focused Imaging (SFI) is newly developed image-enhancing endoscopy technology that enhances the contrast of target tissue structures while improving color contrast because spectral signal energy is further concentrated on the absorption peak wavelength of microvessels by using digital spectral processing techniques. This technology, combined in the latest generation SonoScape's endoscopes (SonoScape Co, Shenzhen, China) with new high-performance LED illumination system, enhances the visibility of colonic mucosal vessels and might increase the detection rate of colorectal polyps. Data available regarding colorectal polyp or adenoma detection with SFI are encouraging but are scanty and limited to back-to back studies.

This two parallel arms, randomized, multicenter trial is aimed at evaluating whether SFI is superior to WLI endoscopy in terms of adenoma detection

DETAILED DESCRIPTION:
45-85 years-old subjects participating in their first colonoscopy and meeting all eligibility criteria are randomised 1:1 to SFI (SFI group) or WLI (WLI group) during insertion and withdrawal phase of colonoscopy. All procedures are performed with a high-definition HD-580 series videocolonscopes with or without magnification (SonoScape Co, Shenzhen, China).

The primary outcome measure is the ADR, defined as the proportion of participants with at least one adenoma (per-patient analysis).

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female aged 45 to 85
* 2. Patients undergoing colonoscopy for the first time due to colorectal cancer screening, having positive fecal immunochemical test (FIT) results, or experiencing gastrointestinal symptoms
* 3. Capable of providing informed consent and agreeing to participate
* 4. Able and willing to follow all research processes

Exclusion Criteria:

* 1. Participated in other clinical trials, signed informed consent form, and in the follow-up period of other clinical trials;
* 2. Participated in clinical trials of drugs and is in the discontinuation period of experimental or control drugs;
* 3. Pregnant or lactating patients;
* 4. Known to have polyposis syndrome;
* 5. Patients with gastrointestinal bleeding;
* 6. Previous history of inflammatory bowel disease, colorectal cancer, or colorectal surgery;
* 7. Patients with contraindications to tissue biopsy;
* 8. History of allergies to the ingredients in intestinal cleansers;
* 9. Individuals with conditions such as intestinal obstruction or perforation, toxic megacolon, heart failure (grade III or IV), severe cardiovascular disease, severe liver failure, or renal insufficiency, among others.
* 10. Researchers believe that patients are not suitable to participate in the trial;
* 11. Have had drug or alcohol abuse or psychological disorders in the past five years.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate (ADR) | 14 days
  ADR was calculated by dividing the total number of patients detected with adenomas by the total number of patients who underwent colonoscopy

SECONDARY OUTCOMES:
Polyp Detection Rate(PDR) | 14 days
  Calculated by dividing the total number of patients with detected polyps by the total number of patients undergoing colonoscopy.
Sessile serrated lesion detection rate (SSLDR) | 14 days
  SSLDR was calculated by dividing the total number of patients detected with sessile serrated lesions by the total number of patients who underwent colonoscopy
Advanced Adenoma Detection Rate | 14 days
  Calculated by dividing the total number of patients with detected advanced adenomas by the total number of patients undergoing colonoscopy.
Mean number of polyps per patient | 14 days
  Calculated by dividing the total number of detected polyps by the total number of patients undergoing colonoscopy.
Mean number of Adenomas per patient(MAP) | 14 days
  Calculated by dividing the total number of detected adenomas by the total number of patients undergoing colonoscopy.
Detection Rate of Polyps of Different Sizes | 14 days
  It is calculated by dividing the number of patients with large (≥10 mm), small (6-9 mm), and diminutive (≤5 mm) polyps by the total number of patients undergoing colonoscopy.
Detection Rate of Adenomas with Different Morphologies | 14 days
  It is calculated by dividing the number of patients with 0-Ip, 0-Is, 0-Isp, and 0-IIa adenomas by the total number of patients undergoing colonoscopy.
Average Number of Adenomas with Different Morphologies | 14 days
  It is calculated by dividing the number of 0-Ip, 0-Is, 0-Isp, and 0-IIa adenomas by the total number of patients undergoing colonoscopy.
Average Number of Polyps of Different Sizes | 14 days
  It is calculated by dividing the number of large (≥10 mm), small (6-9 mm), and diminutive (≤5 mm) polyps by the total number of patients undergoing colonoscopy.
Detection Rate of Adenomas of Different Sizes | 14 days
  It is calculated by dividing the number of patients with large (≥10 mm), small (6-9 mm), and diminutive (≤5 mm) adenomas by the total number of patients undergoing colonoscopy.
Average Number of Adenomas of Different Sizes | 14 days
  It is calculated by dividing the number of large (≥10 mm), small (6-9 mm), and diminutive (≤5 mm) adenomas by the total number of patients undergoing colonoscopy.
Detection Rate of Adenomas in Different Locations | 14 days
  It is calculated by dividing the number of patients with detected adenomas in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon, and cecal region by the total number of patients undergoing colonoscopy.
Average Number of Adenomas in Different Locations | 14 days
  It is calculated by dividing the number of detected adenomas in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon, and cecal region by the total number of patients undergoing colonoscopy.
Detection Rate of Polyps in Different Locations | 14 days
  It is calculated by dividing the number of patients with detected polyps in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon, and cecal region by the total number of patients undergoing colonoscopy.
Average Number of Polyps in Different Locations | 14 days
  It is calculated by dividing the number of detected polyps in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon, and cecal region by the total number of patients undergoing colonoscopy.
Detection Rate of Polyps with Different Morphologies | 14 days
  It is calculated by dividing the number of patients with 0-Ip, 0-Is, 0-Isp, and 0-IIa polyps by the total number of patients undergoing colonoscopy.
Average Number of Polyps with Different Morphologies | 14 days
  It is calculated by dividing the number of 0-Ip, 0-Is, 0-Isp, and 0-IIa polyps by the total number of patients undergoing colonoscopy.
Insertion Time of Colonoscopy | 14 days
  The time taken from the rectum to the cecum.
Withdrawal Time of Colonoscopy | 14 days
  The time taken to complete the examination starting from the cecum.
Cecal Intubation Rate | 14 days
  It is calculated by dividing the number of colonoscopies that reach the cecum by the total number of colonoscopies performed.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Senior Department of Gastroenterology, The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The People'S Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science, Wuhan, Hubei
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - West China School of Public Health West China Fourth Hospital, Chengdu, Sichuan
  - NanChong Center Hospital, Nanchong, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No